CLINICAL TRIAL: NCT07045220
Title: The Effectiveness of a Transtheoretical Model-based Multidisciplinary Collaboration on Cardiac Rehabilitation Outcomes in Patients With Acute Myocardial Infarction：
Brief Title: The Effectiveness of a TTM-based Multidisciplinary Collaboration on Cardiac Rehabilitation Outcomes in Patients With AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhiguo Zou, Doctor, RenJi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Early Myo-TTMCR
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard nursing care and in-hospital CR and routine nursing care was provided for the control group. After clinical assessment, eligible AMI patients received exercise-based in-hospital CR, including lower limb cycle ergometer in bed or on armchair, upper and lower muscle endurance, and 10-60 meters walking. Standard nursing care included patient education on the importance of exercise, suggestions for appropriate exercises based on the disease progression and physiological status, and advises for regular follow-up in the outpatient clinic. After discharge, telephone follow-up was conducted every 1-2 weeks to evaluate the patients' health stat us.
- TTMCR group (Experimental): Patients in the group received a trans-theoretical model (TTM)- based multidisciplinary cardiac rehabilitation program (TTMCR). One day before discharge, physicians, rehabilitation therapists, and nurses jointly developed exercise prescriptions for patients including: exercise frequency, intensity and duration. Nurses and rehabilitation therapists jointly provided patients with cardiac rehabilitation-related health education materials and exercise videos. Physicians recommended that patients use wearable monitoring devices during exercise. After discharge, nurses conducted telephone follow-up once a week for a total of 12 times. The follow-up content mainly included providing sports and medical integration guidance based on the patient's stage of change in exercise behavior.
  Interventions: Behavioral: TTMCR

INTERVENTIONS:
Behavioral: TTMCR — A trans-theoretical model (TTM)- based multidisciplinary CR program (TTMCR) to improve behavior change and cardiac rehabilitation outcomes
  Arms: TTMCR group

SUMMARY:
Cardiac rehabilitation (CR) has been shown to reduce morbidity and mortality in patients with acute myocardial infarction (AMI), however, the proportion of patients participating in and benefiting from cardiac rehabilitation (CR) remains low in China. This study aims to explore the effects of a trans-theoretical model (TTM)- based multidisciplinary CR program (TTMCR) on behavior change and CR outcomes in AMI patients.

DETAILED DESCRIPTION:
We recruited 86 eligible patients hospitalized with AMI were enrolled from a tertiary hospital and allocated into two groups: the intervention group (TTMCR group, n = 43) received TTM-based behavioral stage-matched education, individualized exercise prescription, and ongoing support via a multidisciplinary care team consisting of physicians, nurses, rehabilitation therapists, and cardiac rehabilitation specialists. The control group (n = 41) received standard nursing care and in-hospital CR education without structured follow-up.

The intervention lasted 12 weeks and included pre-discharge assessment and education, individualized home-based exercise prescriptions, telephone follow-ups, social media-based communication (WeChat), and outpatient online consultation support. Outcome measures were assessed at baseline and at 3 months post-discharge. The primary outcomes included objective cardiopulmonary function parameters measured by cardiopulmonary exercise testing (CPET)-specifically anaerobic threshold oxygen consumption per kilogram (AT-VO2/kg) and peak oxygen consumption per kilogram (VO2 Peak/kg)-as well as subjective measures including the Exercise Self-Efficacy Scale (ESES) and the Exercise Social Support Scale (ESSS). The secondary outcome was behavioral change, assessed by weekly exercise frequency and the Stages of Exercise Behavior Change Scale.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years old;
* Diagnosed with AMI according to the European Society of Cardiology (ESC) guidelines;
* Received standard PCI and drug treatment in the hospital;
* Able to communicate effectively with healthcare providers in Mandarin;
* Long-term residents of Shanghai who had been living in Shanghai for at least 6 months prior to the study and intended to continue residing in Shanghai for the duration of the intervention and follow-up period (3 months);
* Voluntary participation in the study with signed informed consent;

Exclusion Criteria:

* Contraindications to cardiac rehabilitation;
* History of mental disorders;
* Withdrawal from the study for any reason;
* Participating in other intervention research projects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
3-month change in VO2 Peak-/kg | VO2 Peak-/kg of each patient was assessed by CPET at baseline and at 3-month follow-up.
  Peak ventilation oxygen per kilogram (VO2 Peak-/kg) reflects the patient's exercise capacity and is an important measurement parameter in cardiopulmonary exercise testing (CPET). In this study, 3-month change of VO2 Peak-/kg was used to assess the outcomes of cardiac rehabilitation.
3-month change in AT-VO2/kg | AT-VO2/kg of each patient was assessed by CPET at baseline and at 3-month follow-up.
  Ventilation oxygen at the anaerobic threshold per kilogram (AT-VO2/kg ) reflects the patient's exercise capacity and is an important measurement parameter in CPET. In this study, 3-month change of AT-VO2/kg was used to assess the outcomes of cardiac rehabilitation.
3-month change of ESES score | ESES score of each patient was assessed at baseline and at 3-month follow-up.
  Exercise Self-Efficacy Scale (ESES) was developed to developed by to assess patients' confidence in the ability to participate in exercise and overcome difficulties during exercise. In this study, the ESES score was used as a subjective index to assess the outcomes of cardiac rehabilitation.
3-month change of ESSS scores | ESSS score of each patient was assessed at baseline and at 3-month follow-up.
  Exercise Social Support Scale (ESSS) is a tool used to assess the level of social support individuals perceive related to their exercise habits. In this study, the ESSS score was used as a subjective index to assess the outcomes of cardiac rehabilitation.

SECONDARY OUTCOMES:
Weekly exercise frequency | Weekly exercise frequency was assessed at baseline and at 3-month follow-up.
  Weekly exercise frequency refers to the number of times a patient engages in structured physical activity (aerobic or resistance exercise) lasting at least 30 minutes per session, within a 7-day period. In this study, the change in weekly exercise frequency was evaluated to determine the effects of treatments on behavior change.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No